CLINICAL TRIAL: NCT04245930
Title: A Randomized and Controlled Study of Efficacy and Safety of Bovine Pericardial Patch and TiLOOP® Bra Mesh in Patients With Immediate Implant Breast Reconstruction.
Brief Title: Bovine Pericardial Patch and TiLOOP® Bra Mesh in Immediate Implant Breast Reconstruction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2019453
Record Dates: First submitted 2020-01-28; First posted 2020-01-29 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Implant Breast Reconstruction; TiLOOP® Bra Mesh; Bovine Pericardial Patch

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bovine Pericardial Patch (Active Comparator): Immediate implant breast reconstruction using bovine pericardial patch. n=88
  Interventions: Procedure: Bovine Pericardial Patch in Immediate Implant Breast Reconstruction
- TiLOOP® Bra Mesh (Experimental): Immediate implant breast reconstruction using TiLOOP® Bra Mesh. n=88
  Interventions: Procedure: TiLOOP® Bra Mesh in Immediate Implant Breast Reconstruction

INTERVENTIONS:
Procedure: Bovine Pericardial Patch in Immediate Implant Breast Reconstruction — Patients will receive immediate breast implant reconstruction using Bovine Pericardial Patch
  Arms: Bovine Pericardial Patch
Procedure: TiLOOP® Bra Mesh in Immediate Implant Breast Reconstruction — Patients will receive immediate breast implant reconstruction using TiLOOP® Bra Mesh
  Arms: TiLOOP® Bra Mesh

SUMMARY:
This study is the first randomized and controlled study assessing the efficacy and safety of bovine pericardial patch and TiLOOP® bra mesh in patients with immediate implant breast reconstruction

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with I~II stage breast cancer and Intent to receive NSM or SSM and implant based breast reconstruction
2. Do not smoking in the last 4 weeks or more
3. Mental health patients
4. Signed consent to participate

Exclusion Criteria:

1. Locally advanced stage patients or patients with distal metastasis
2. Patients received thoracic wall radiotherapy or will receive radiotherapy
3. Smoking in the last 4 weeks
4. Anticipated implant volume more than 600cc
5. Patients of pregnancy or lactation
6. Patients received neoadjuvant therapy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Complication Rates | up to 12 months after surgery
  The rate of complications in the two groups

SECONDARY OUTCOMES:
Patient satisfaction-Breast-Q questionnaire | up to 12 months after surgery
  We use the Breast-Q questionnaire to evaluate patients' satisfaction via the reconstruction module of BREAST-Q.
Cosmetic outcome of reconstructed breast | Immediately, up to 3 months, 6 months and 12 months after surgery
  Harris evaluation score was used to evaluate the aesthetic outcome of patients' reconstructed breasts, which was scored as "excellent," "good," "fair," "poor".
The rate of surgical revision of reconstructed breasts | up to 12 months after surgery
  To record the rate of surgical revision events of the reconstructed breasts
Health economics-inpatient cost | up to 12 months after surgery, including the cost of surgical revision
  Hospital inpatient costs due to immediate implant breast reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Jian Yin, MD., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided